CLINICAL TRIAL: NCT05625256
Title: Clinical Validation of the SentiCor-300 Continuous Noninvasive Blood Pressure Against Invasive Arterial Blood Pressure
Brief Title: Validation of the SentiCor-300 Continuous Noninvasive Blood Pressure
Status: Withdrawn | Type: Observational
Why Stopped: Funding
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 22-511
Record Dates: First submitted 2022-11-06; First posted 2022-11-22 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Blood Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Accuracy of Continuous Noninvasive Blood Pressure at Various Stages of Anesthesia: To compare noninvasive continuous arterial pressures obtained from the SentiCor-300 with direct intra-arterial blood pressure measurements at various stages of anesthesia (such as induction, laryngoscopy, maintenance, emergence, and recovery) and after emergence in various positions.
  Interventions: Device: SentiCor-300

INTERVENTIONS:
Device: SentiCor-300 — Continuous blood pressure measurement with the SentiCor-300.

SUMMARY:
To compare continuous arterial pressures obtained from the SentiCor-300 with direct intra-arterial blood pressure measurements at various stages of anesthesia (such as induction, laryngoscopy, maintenance, emergence, and recovery) and after emergence in supine position.

DETAILED DESCRIPTION:
Analysis of number and magnitude of BP changes Adjust endpoint calculation definitions and methods based on this lead in results Estimate sample size for main study Demonstration of capability to quantify and annotate interference in the arterial line signal and detect and changes in patient orientation Parallel recording of SentiCor-300 PPG sensor

Main study:

Validate SentiCor-300 noninvasive blood pressure against direct arterial pressure measurements.

Up to 200 (10 run-in, the balance- study) Run in phase will be performed with Senticor-100, data will be used for sample size estimation of balance study.

ELIGIBILITY:
Inclusion Criteria:

* Clinical indication for arterial catheter insertion;
* Age ≥18 years;
* American Society of Anesthesiologists (ASA) physical status class ≤3;
* Enrollment will be adjusted as necessary so the final population includes at least 40% men and 40% women;
* Planned length of surgery >60 minutes;
* Anticipated supine positioning;
* Anticipated initial recovery in the post-anesthesia care unit.

Exclusion criteria:

* Severe peripheral vascular disease;
* Surgery that involves manipulation of large arteries
* Bypass surgery
* Positive Allen's test
* Inability to insert a catheter into an upper extremity artery;
* Patients with an arterial-venous shunt for hemodialysis;
* Inability to measure NIBP on the arm with the arterial catheter;
* Atria l fibrillation;
* Body Mass Index (BMI) >35kg/m2;
* Esophageal or nasopharyngeal pathology, coarctation of the aorta;
* Emergency surgery.
* Surgery which involves manipulation of major arteries

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consenting adults scheduled for elective major surgery that requires an arterial catheter will be recruited into the study. There will be no restriction on race or ethnicity.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-06 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Accuracy | During hospital admission
  The difference between SentiCor-300 and the actual intra-arterial blood pressure for systolic and diastolic pressures.

SECONDARY OUTCOMES:
Change | During hospital admission
  Comparison of continuous arterial pressures obtained from the SentiCor-300 with direct intra-arterial blood pressure measurements during hemodynamic changes at various stages of anesthesia (such as induction, laryngoscopy, maintenance, emergence, and recovery) and after emergence in various postures and positions.
Calibration Duration | During hospital admission
  To determine how long an oscillometric calibration of the SentiCor-300 lasts.
Gender and Fitzpatrick index | During hospital admission
  To compare perform class analysis on accuracy versus gender and Fitzpatrick index.

CONTACTS AND LOCATIONS:
Overall Officials: Alparslan Turan, MD, Principal Investigator — The Cleveland Clinic

IPD SHARING:
Plan to Share IPD: No